CLINICAL TRIAL: NCT00774059
Title: Phase 1 Study to Evaluate the Safety and Performance of the Orbix Breast Lift System
Brief Title: Evaluation of Safety and Performance of the Orbix Breast Lift System
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No EC approval obtained
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Adi Cohen, Orbix Medical
Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC 08-1-024
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Breast Ptosis
Keywords: Breast ptosis, Breast lift

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: Breast lift system — During a breast operation for ptosis a device is brought into the breast and attached to the ribs, to provide lifting of the breast

SUMMARY:
The study is using a new breast lift system to complement a breast-lift operation.

In general there will be recurrence of breast-ptosis after a correcting operation.

With this device we want to minimize this recurrence and provide an "internal bra".

ELIGIBILITY:
Inclusion Criteria:

1.Female subject between 30-50 years of age 2. Subject is referred for mastopexy(breast lifting)due to one of the following reasons:

* Breast ptosis grade I or II (minimal invasive)
* Breast ptosis grade I to IV (open procedure)
* pseudoptosis following breast reduction surgery 3. subject willing to participate as evidenced by signing the written informed consent 4. Minimal invasive: breast cup size <C

Exclusion Criteria:

1. Pregnant or lactating women
2. history of surgical procedures involving the ribs and rib cage
3. Osteoporosis
4. breast implants
5. breast carcinoma
6. auto-immune disease -

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Result after using the breast lift system,recurrence of ptosis. | one year

SECONDARY OUTCOMES:
complications | one year

CONTACTS AND LOCATIONS:
Overall Officials: Marjoes MP Schuckman, MD, Principal Investigator — Maastricht University Hospital; Adi Cohen, Study Director — Orbix medical
Locations (1):
- Maastricht Univeristy Hospital, Maastricht, Netherlands